CLINICAL TRIAL: NCT05164393
Title: A Single-center, Randomized Double-blind, Vehicle-controlled, Dose-ranging Decentralised Clinical Trial to Evaluate the Safety and Efficacy of Daily Field-directed Topical Applications of AVX001 Silicone-based Gel in Doses of 1% or 3% in Adult Subjects With Multiple Actinic Keratosis Lesions Olsen Grade 1 or 2
Brief Title: Phase I/IIa Trial to Evaluate AVX001 Gel in Doses of 1% or 3% Compared With Vehicle Over Four Weeks of Field-directed Treatment Period in Adult Subjects With AK
Acronym: COAKS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Coegin Pharma AB (Industry)
Collaborators: Studies&Me (Industry); Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVXCLIN005; 2021-000934-32 (EudraCT Number)
Record Dates: First submitted 2021-11-22; First posted 2021-12-20 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Actinic Keratoses
Keywords: Actinic Keratosis; Olsen grade; Actinic Keratosis Field Assessment Scale; Local skin reaction; Topical treatment
MeSH Terms: conditions — Keratosis, Actinic | interventions — AVX001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AVX001 1% (Experimental): Application of AVX001 1% gel to treatment field once daily
  Interventions: Drug: AVX001
- AVX001 3% (Experimental): Application of AVX001 3% gel to treatment field once daily.
  Interventions: Drug: AVX001
- AVX001 Vehicle (Placebo Comparator): Application of AVX001 vehicle gel to treatment field once daily
  Interventions: Drug: AVX001

INTERVENTIONS:
Drug: AVX001 — Topical gel treatment for once daily application

SUMMARY:
Actinic keratosis (AK), also known as solar keratosis, is a common skin condition characterised by abnormal growth of skin cells caused by long-term sun exposure. AK is considered to be a precancerous lesion, and is therefore commonly treated to reduce the risk of malignant transformation into skin cancer.

The trial is a randomised, double-blind, vehicle-controlled, dose-comparison trial in which adult subjects with AK grade 1 or 2 will be treated with AVX001 silicone-based gel in doses of 1% or 3% or with a gel vehicle for a 4-week field-directed treatment period. Subjects will be followed up for 8 weeks after the treatment period. The primary objective is to evaluate the local tolerability of daily applications of AVX001 gel in doses of 1% or 3% and compare with vehicle.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent
2. ≥ 18 years of age
3. Fluent in Danish
4. Clinical AK diagnosis confirmed by PI.
5. Present an area of 25cm2 with 4 to 8 AK lesions located in face, neck or chest AK lesions in target area severity grade 1 or 2 as defined by the Olsen clinical Criteria for AK
6. Able to and willing to follow trial procedures including application of AVX001 and using the Study App.
7. Have a suitable smartphone to complete the trial tasks (Android operating system: Android 8.1 or higher; iPhone with iOS 12.4 or higher)
8. Female subjects must either be of non-childbearing potential (either be surgically sterile (hysterectomy or tubal ligation) or post-menopausal) or must be using a highly effective method of contraception. Contraception must be maintained for the duration of the study.

   * A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
   * A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient. (CTFG 2020)
   * For women not taking hormonal contraception with amenorrhea for less than 12 months and just a single FSH measurement in postmenopausal range, a decision can be made by the PI whether it is appropriate for them to undergo a confirmatory FSH measurement or commence a highly effective method of birth control
   * Highly effective methods of birth control are defined as those, alone or in combination, that result in a low failure rate (less than 1% per year) when used consistently and correctly. (ICH 2009)

Such methods include:

* Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation : oral, intravaginal, transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system ( IUS)
* Bilateral tubal occlusion
* Vasectomised partner.
* Sexual abstinence.

Exclusion Criteria:

1. AK lesions classified as Olsen grade 3 in target area
2. Atypical AK lesions in the target area, including suspected SCC or BCC
3. Under suspicion of, or current skin cancer diagnosis in the target area. subjects who had BCC, SCC or melanoma and have completed curative therapy at least 12 months prior to screening and are in remission can be considered to participate in the trial by investigator's discretion
4. Any dermatological condition in the target area that can be exacerbated by treatment or affect trial assessments, including but not limited to psoriasis vulgaris AD, rosacea, urticaria, scabies, and herpes simplex
5. Received immunosuppressive/immunomodulating drugs including but not limited to methotrexate, cyclosporine, azathioprine, oral retinoids, 6 months prior to baseline visit.
6. Received systemic corticosteroids including but not limited to betamethasone, prednisone, dexamethasone, methylprednisolone (except if via inhale or intranasal delivery) 6 months prior to baseline visit.
7. Received lesion or field directed therapy within 2 cm of the target area for trial treatment one month prior to baseline visit, including topical drugs, including but not limited to

   * topical fluorouracil, imiquimod, ingenol mebutate and diclofenac.
   * destructive therapies, including but not limited to surgery, cryotherapy, dermabrasion, and photodynamic therapy
   * field ablation treatments, including but not limited to chemical peels, laser resurfacing
8. Recipient of organ transplant including but not limited to bone marrow, kidney, liver, heart
9. Any unstable neurological or psychiatric disorder based on the investigator's opinion which has the potential to affect the safety of the subject, influence on trial objectives or impede the subject's ability to complete the trial.
10. History of chronic alcohol or drug abuse within 12 months prior to screening or any condition associated with poor compliance at the investigator's discretion
11. Received treatment with any non-approved drug substance within the last 4 weeks prior to baseline visit.
12. Known allergy or intolerance to fish, shellfish or fish oil
13. Concurrent participation in any other clinical trial or participation in any clinical trial treatments 4 weeks prior to enrolment.
14. Subject is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with local skin reaction (LSR) >2 | Baseline to end of study (12 weeks)

SECONDARY OUTCOMES:
Assessment of safety based on frequency of SAEs | Baseline to end of study (12 weeks)
Assessment of safety based on frequency of AEs | Baseline to end of study (12 weeks)
Assessment of safety based on skin examinations | Baseline to end of study (12 weeks)
Assessment of safety based on blood pressure (vital sign) | Baseline to end of study (12 weeks)
Assessment of safety based on pulse (vital sign) | Baseline to end of study (12 weeks)
Assessment of safety based on temperature (vital sign) | Baseline to end of study (12 weeks)
Proportion of subjects who experience LSR grade 1, 2, 3 and 4 | Baseline to End of Treatment and End of Study (week 4)
Proportion of subjects experiencing a clinically visible clearance of target area of >50% as assessed in-clinic | Baseline to the end of treatment visit (EOT) (week 4) / early termination.
Proportion of subjects experiencing a clinically visible clearance of target area of >50% as assessed in-clinic | Baseline to the end of the study visit (EOS, week 12).
Recurrence rate of AKs as assessed in-clinic after treatment clearance | Between End of Treatment (week 4) and End of Study visits (week 12).
Appearance of new lesions in the target area as assessed in-clinic | From Baseline to EOS (week 12)
Subject satisfaction with the AVX001 gel, assessed by TSQM | at Week 2 and EOT (week 4).
Proportion of patients with a cosmetic outcome grade <2 , as assessed using the Cosmetic Scoring Tool. | from Baseline to EOS (week 12)
Cosmetic outcome of target area as evaluated by participants by comparing the status at EOS with a baseline photo | Baseline and End of Study (week 12)

OTHER OUTCOMES:
Changes in AK-FAS , as evaluated by the Central Assessors on the smartphone photos taken by the subjects. | From Baseline to EOT and EOS
The level of agreement between AK-FAS in-clinic, and AK-FAS performed remotely by Central Assessors using smartphone photos taken by the subjects | From Baseline to End of Study
Proportion of subjects presenting with an LSR>2, as evaluated by the Central Assessors on the smartphone photos taken by the subjects | from Baseline to EOT, and EOS
Proportion of subjects who experience LSR grade 1, 2, 3 and 4, as evaluated by the Central Assessors on the smartphone photos taken by the subjects | from Baseline to EOS
Time to reach a clinically visible clearance of target area of >50% for all enrolled subjects performed from remote by Central Assessors using smartphone photos taken by the subjects. | From Baseline to End of Study
Presence of AK-related skin changes evaluated by non-invasive optical imaging | At baseline and EOS

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD, PhD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ortner VK, Johansen B, Kilov K, Castillo Mondragon A, Duvold T, Kihl J, Ashcroft FJ, Feuerherm AJ, Pind Laugesen C, Marcker Espersen ML, Manole I, Isberg AP, Andersen AD, Rakvaag E, Zibert JR, Haedersdal M. The Copenhagen Actinic Keratosis Study (COAKS). A decentralised clinical trial to evaluate tolerability, safety and efficacy of daily field-directed topical treatment with cytosolic phospholipase A2 inhibitor, AVX001, in participants with actinic keratosis: protocol for a randomised controlled phase I/IIa trial. BMJ Open. 2022 Oct 5;12(10):e061012. doi: 10.1136/bmjopen-2022-061012. PMID 36198452